CLINICAL TRIAL: NCT05492175
Title: Proximal- Versus Distal-Prioritized Robotic Practice Plus Kinetic Exergaming in Stroke Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-M-161
Record Dates: First submitted 2022-07-03; First posted 2022-08-08 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Stroke Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- proximal-prioritized robotic practice plus kinetic exergaming group (Experimental): 60 minutes per day, 3 days per week for 6 weeks
  Interventions: Other: robotic practice; Other: kinetic exergaming
- distal-prioritized robotic practice plus kinetic exergaming group (Active Comparator): 60 minutes per day, 3 days per week for 6 weeks
  Interventions: Other: robotic practice; Other: kinetic exergaming
- robotic practice plus conventional therapy group (Active Comparator): 60 minutes per day, 3 days per week for 6 weeks
  Interventions: Other: robotic practice; Other: conventional therapy

INTERVENTIONS:
Other: robotic practice — According to the group assignment, participants will start from the BMT proximal mode (i.e., forearm pronation-supination movement), and then the distal mode (i.e., wrist flexion-extension movement), and vice versa. Each participant is expected to complete approximately 400 to 600 repetitions of the proximal mode session (i.e., forearm movements) and another 400 to 600 repetitions of the distal mode session (i.e., wrist movements), respectively.
Other: kinetic exergaming — All of the participants in experimental and comparison groups will practice on the exergaming for 30 minutes per session. To avoid fatigue, the four domains of programs will be provided alternately. Each program will be executed for approximately 5 minutes with warm-up, followed by a 2-minute break between programs, and cool-down. The games will be selected and adapted according to the personal capacity, the occupational role, and the rehabilitation goal of each participant. The investigators will illustrate and guide the participants to play the games and stand next to them to prevent falls from occurring. To increase security, we will place a handrail in front of the participant for support as needed.
  Arms: distal-prioritized robotic practice plus kinetic exergaming group; proximal-prioritized robotic practice plus kinetic exergaming group
Other: conventional therapy — Participants in control group will receive 30 minutes of therapist-mediated conventional therapy per session. The training protocols of the conventional therapy will use occupational therapy techniques, such as neurodevelopmental techniques and functional task training. The therapy will be adapted to the participants' levels of motor deficits and their personal needs. The protocol will include affected arm exercise or gross motor training, muscle strengthening of the affected arm, fine motor or dexterity training, and functional tasks of daily life or compensatory techniques to alleviate functional deficits. The content of the functional tasks will be decided together by participants and therapists, such as picking up and putting down items in a box, lifting two soft drink bottles, and so on.
  Arms: robotic practice plus conventional therapy group

SUMMARY:
This research program aims at investigating the effects of upper-limb robotic therapy primed with interactive exergaming as an innovative hybrid regimen in stroke rehabilitation.

DETAILED DESCRIPTION:
Robotic therapy can potentially be a movement-based priming technique to promote rebalancing of cortical excitability and create an enriched neuroplastic environment by priming the brain to facilitate motor and functional recovery. The proximal priority and distal priority robotic priming techniques may bring differential effects. This proposed research project aims to: (1) examine the effects of proximal priority versus distal priority of bilateral robotic priming combined with exergaming on sensorimotor function, daily function, self-efficacy, quality of life, and motor control strategy in patients with stroke, (2) investigate the 3-month retention effects of the three approaches, and (3) identify the potential predictors of functionally relevant changes after therapy.

ELIGIBILITY:
Inclusion Criteria:

1. a first ever-stroke≧3 months
2. age range between 20 to 80 years
3. baseline Fugl-Meyer assessment of upper extremity scale (FMA-UE) between 18 to 56
4. no excessive muscle spasticity of the affected extremities (Modified Ashworth Scale < 3 at any joints)
5. able to follow examiners' commands and study instructions (Mini-Mental State Examination score≧22)
6. can maintain a step-standing position for at least 30 seconds
7. can walk for at least 10 meters with or without device
8. no participation in further experimental rehabilitation or drug studies during the duration of the project

Exclusion Criteria:

1. acute inflammation and pain
2. concomitant neurologic, neuromuscular or orthopedic conditions that may impede participation in this research.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Fugl-Meyer Assessment (FMA) at 6 weeks and 18 weeks | Baseline, 6 weeks, and 18 weeks
  1. The upper-extremity subscale of the FMA will be used to assess motor impairment.
  2. There are 33 UE items that assess movements and reflexes of the shoulder/elbow/forearm, wrist, and hand, and coordination/speed. Each item is on a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully).
  3. The maximum score is 66, with a subscale score of 42 for the proximal part of the arms (shoulder/elbow) and 24 for the distal part of the arm (wrist/hand/coordination)
  4. The higher summed score means the greater recovery of motor impairment.
Change from Baseline 10 meter walk test (10-MWT) at 6 weeks and 18 weeks | Baseline, 6 weeks, and 18 weeks
  1.10 meter walk test is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.
  2.The total time is recorded in m/s 3.The lower total time means the greater recovery of walking speed.

SECONDARY OUTCOMES:
Medical Research Council scale (MRC) | Baseline, 6 weeks, and 18 weeks
  1. MRC measures muscle power of the affected arm and is scored on a 6-point ordinal scale (0 = no contraction, 5 = resisted to maximal strength, full power compared with the unaffected side)
  2. The higher score means the greater muscle power.
The ActiGraph GX3 accelerometers (ActiGraph, Shalimar, FL,USA) | Baseline, 6 weeks, and 18 weeks
  1. Accelerometry is used to measure human movement. These devices record patterns of motion and non-motion.
  2. All participants will be asked to wear the devices for 3 consecutive days before and after the intervention.
  3. .The accelerometer will record the number of movements per minute, and the mean counts of movements per minute will be calculated.
  4. The higher mean counts of movements per minute means the more activity of arm.
Functional Independence Measure (FIM) | Baseline, 6 weeks, and 18 weeks
  1. The FIM consists of 18 items grouped into 6 sub-scales, including self-care, sphincter control, transfer, locomotion, communication, and social cognition.
  2. Each item is rated from 1 (full assistance) to 7 (full independence), according to the level of support required to perform the tasks.
  3. A higher score (maximum score of 126) indicates a lower disability.
Stroke Self-Efficacy Questionnaire (SSEQ) | Baseline, 6 weeks, and 18 weeks
  1. The SSEQ will be used to gauge participants' confidence in their functional performance after stroke.
  2. It includes 13 items and gives an overview of the factors that influence functional performance.
  3. Each item will be assigned according to the perceived confidence rating on the scale of 0 (no confidence at all) to 10 (full confidence).
  4. The higher summed score means the more confidence of participant.
Adverse events (pain and fatigue) | through study completion, an average of 18 weeks
  1. Self-reported fatigue and pain severity will be evaluated using the 10-cm vertical line in the Face Rating Scale for adverse effects.
  2. The participants will rate the level of their pain and fatigue after the intervention on an 11-point ordinal scale (0 = no pain/fatigue; 10 = the most severe pain/fatigue).
  3. The higher score means the more pain or fatigue of participant.

CONTACTS AND LOCATIONS:
Overall Officials: Keh-Chung Lin, Sc.D, Principal Investigator — National Taiwan University
Locations (4):
- Taiwan (4):
  - Feng Yuan Hospital, Ministry of Health and Welfare, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Municipal Wan Fang Hospital, Taipei
  - Taipei Tzu Chi Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No